CLINICAL TRIAL: NCT07223203
Title: TRITON-PN: A Phase 3, Global, Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Nucresiran in Patients With Hereditary Transthyretin-Mediated Amyloidosis With Polyneuropathy (hATTR-PN)
Brief Title: TRITON-PN: A Study to Evaluate the Efficacy and Safety of Nucresiran in Patients With Hereditary Transthyretin Amyloidosis With Polyneuropathy
Acronym: TRITON-PN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTRSC04-004; 2025-522544-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Transthyretin-Mediated Amyloidosis With Polyneuropathy; hATTR-PN
Keywords: Polyneuropathy; Amyloidosis; Transthyretin; TTR; RNAi therapeutic
MeSH Terms: conditions — Polyneuropathies; Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nucresiran 300 mg (Experimental): Patients will be administered nucresiran 300 mg subcutaneously (SC) once every 6 months (q6M) during the Treatment Period and Treatment Extension Period
  Interventions: Drug: Nucresiran
- Vutrisiran 25 mg followed by Nucresiran 300 mg (Active Comparator): Patients will be administered vutrisiran 25 mg SC every 3 months (q3M) during the Treatment Period followed by nucresiran 300 mg SC q6M during the Treatment Extension Period
  Interventions: Drug: Nucresiran; Drug: Vutrisiran

INTERVENTIONS:
Drug: Nucresiran — Nucresiran 300 mg administered SC q6M
  Other Names: ALN-TTRSC04
Drug: Vutrisiran — Vutrisiran 25 mg administered SC q3M
  Other Names: AMVUTTRA; ALN-TTRSC02
  Arms: Vutrisiran 25 mg followed by Nucresiran 300 mg

SUMMARY:
The purpose of this study is to:

* Determine the efficacy of nucresiran in patients with hATTR-PN by evaluating the effect on neurologic impairment, quality of life, nutritional status, disability, and gait speed
* Demonstrate superiority of nucresiran compared to in-study vutrisiran with respect to serum transthyretin (TTR) levels

ELIGIBILITY:
Inclusion Criteria:

* Has documented diagnosis of hATTR-PN
* Has a diagnosis of hATTR amyloidosis with polyneuropathy with a documented TTR gene variant
* Has a neuropathy impairment score (NIS) of 5 to 130 (inclusive)
* Has a Karnofsky Performance Status (KPS) of ≥60%

Exclusion Criteria:

* Has had a liver transplant or is likely, in the opinion of the Investigator, to undergo liver transplantation during the Treatment Period of the study
* Has known other (non-hATTR) forms of amyloidosis or clinical evidence of leptomeningeal amyloidosis
* Has a New York Heart Association (NYHA) heart failure classification >2
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 upper limit of normal (ULN)
* Has total bilirubin >1.5 ULN
* Has estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73m^2
* Has other known causes of sensorimotor or autonomic neuropathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2027-12-27 (Estimated); Study Completion 2031-06-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Modified Neuropathy Impairment Score +7 (mNIS+7) Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 9 | Baseline and Month 9
  The mNIS+7 is a composite score that measures neurologic impairment which includes the following components: physical exam of lower limbs, upper limbs and cranial nerves to assess motor strength/weakness and deep tendon reflexes, electrophysiologic measurement of large nerve fiber function, sensory testing and postural blood pressure. The mNIS+7 is scored from 0 (no impairment) to 304 points (maximum impairment). A higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Change from Baseline in Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QoL-DN) Total Score Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 9 | Baseline and Month 9
  The Norfolk QoL-DN is a standardized 35-item patient-rated questionnaire used to assess 5 domains: physical function, large fiber neuropathy, activities of daily living, symptoms, small fiber neuropathy, and autonomic neuropathy. The minimum and maximum values are -4 and 136, respectively. A higher score indicates a worse outcome.
Percent Reduction in Serum TTR Levels in the Nucresiran Group Compared to the In-study Vutrisiran Group through Month 9 | Up to Month 9
Change from Baseline in Modified Body Mass Index (mBMI) Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 9 | Baseline and Month 9
  The mBMI, which is a measure of nutritional status, is calculated as the product of body mass index (BMI) (weight in kilograms divided by the square of height in meters) and serum albumin (g/L) to reflect fluid balance, such as fluid accumulation or dehydration. A negative change from baseline indicates a better outcome.
Change from Baseline in the mNIS+7 Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 18 | Baseline and Month 18
  The mNIS+7 is a composite score that measures neurologic impairment which includes the following components: physical exam of lower limbs, upper limbs and cranial nerves to assess motor strength/weakness and deep tendon reflexes, electrophysiologic measurement of large nerve fiber function, sensory testing and postural blood pressure. The mNIS+7 is scored from 0 (no impairment) to 304 points (maximum impairment). A higher score indicates a worse outcome.
Change from Baseline in Norfolk QoL-DN Total Score Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 18 | Baseline and Month 18
  The Norfolk QoL-DN is a standardized 35-item patient-rated questionnaire used to assess 5 domains: physical function, large fiber neuropathy, activities of daily living, symptoms, small fiber neuropathy, and autonomic neuropathy. The minimum and maximum values are -4 and 136, respectively. A higher score indicates a worse outcome.
Change from Baseline in mBMI Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 18 | Baseline and Month 18
  The mBMI, which is a measure of nutritional status, is calculated as the product of body mass index (BMI) (weight in kilograms divided by the square of height in meters) and serum albumin (g/L) to reflect fluid balance, such as fluid accumulation or dehydration. A negative change from baseline indicates a better outcome.
Change from Baseline in Rasch-built Overall Disability Scale (R-ODS) Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 18 | Baseline and Month 18
  The R-ODS is a patient-reported measure of level of disability on a scale of 0-48, with 0 being the worst and 48 the best (no limitations); scores are based on activities of daily living and social participation. An increase in R-ODS from baseline suggests improvement in disability, and a decrease from baseline suggests worsening of disability.
Change from Baseline in Timed 10-meter Walk Test (10-MWT) Compared to the External Placebo Group from the APOLLO Study (NCT01960348) at Month 18 | Baseline and Month 18
  The timed 10-MWT is a measure of ambulatory ability and measures the time (in seconds) that it takes a participant to walk 10 meters (gait speed). An increase in gait speed from baseline represents improvement, and a decrease from baseline represents worsening.
Percent Reduction in Serum TTR Levels in the Nucresiran Group Compared to the In-study Vutrisiran Group through Month 18 | Up to Month 18
Percent Reduction in Serum TTR Levels in the Nucresiran Group Compared to the In-study Vutrisiran Group at Week 6 | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals Inc
Locations (1):
- Clinical Trial Site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Phase 2-4 trials:
  Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.